CLINICAL TRIAL: NCT03175029
Title: Exploratory Study of TAC-302 in Detrusor Underactivity Patients With Overactive Bladder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10054040
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Detrusor Underactivity; Overactive Bladder
Keywords: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Bladder, Underactive; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms | interventions — tac-302

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAC-302 (Experimental)
  Interventions: Drug: TAC-302
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAC-302 — TAC-302 200 mg administered orally twice per day after meals, for 12 weeks.
  Arms: TAC-302
Drug: Placebo — Placebo administered orally twice per day after meals, for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAC-302 in detrusor underactivity patients with overactive bladder.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of TAC-302 for 12 weeks in detrusor underactivity patients with overactive bladder by measuring the following parameters of pressure-flow study.

* Male; bladder contractility index (BCI)
* Female; projected isovolumetric pressure (PIP) 1

ELIGIBILITY:
Key Inclusion Criteria:

* To have Lower Urinary Tract Symptoms for at least 12 weeks prior to study entry
* To have at least 1 urinary urgency episodes per day, and diurnal urinary frequency of 8 or more per day.
* To meet the detrusor underactivity criteria by urodynamic study

Key Exclusion Criteria:

* Neurogenic bladder by the central nervous system diseases.
* StageIII or more cystocele of pelvic organ prolapse quantification system (women)
* Prostate volume ≥30mL (Men)
* Any symptoms of Urinary tract infection (UTI)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd, Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- Taiho Pharmaceutical Co., Ltd selected site, Kumamoto, Japan

REFERENCES:
- [Derived] Yoshida M, Gotoh M, Yokoyama O, Kakizaki H, Yamanishi T, Yamaguchi O. Efficacy of TAC-302 for patients with detrusor underactivity and overactive bladder: a randomized, double-blind, placebo-controlled phase 2 study. World J Urol. 2022 Nov;40(11):2799-2805. doi: 10.1007/s00345-022-04163-4. Epub 2022 Oct 7. PMID 36205739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 21 medical institutions in Japan and the study period was from September 9, 2017 to November 14, 2019.
  Of the 213 patients who gave informed consent and received screening tests, 18 patients were withdrawn at screening. The number of patients enrolled in the observation period was 195 patients, but after the end of the observation period, 76 patients were determined to be eligible for enrollment in the treatment period.
Period: Overall Study
Arm/Group | TAC-302 | Placebo
Started (Full analysis set (FAS) was used for the analysis. FAS included all patients who took the study drug at least once and had at least one efficacy measurement before and during the treatment period.) | 52 | 24
Completed | 49 | 23
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Study treatment becomes impossible due to changing hospital or other reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol set (PPS) was used for the analysis. PPS included all patients in the Full analysis set (FAS) with no inclusion/exclusion criteria violations, who were compliant for ≥ 80% of the treatment period, were not administered any prohibited concomitant medication or therapy during the study period, and had a week 12 evaluation of the primary endpoint. FAS included all patients who took the study drug at least once and had ≥ 1 efficacy measurement before and during the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAC-302 | Placebo | Total
Number analyzed (Participants) | 42 | 18 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (10.7) | 70.4 (9.1) | 70.8 (10.2)
Age, Continuous [Median (Full Range); unit: years] | 74.0 [46 to 90] | 73.5 [44 to 84] | 74.0 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 27 | 11 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 42 | 18 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Duration of lower urinary tract symptoms [Mean (Standard Deviation); unit: months] | 92.2 (95.1) | 72.9 (71.1) | 86.4 (88.4)
Duration of lower urinary tract symptoms [Median (Full Range); unit: months] | 79.0 [4 to 483] | 45.5 [12 to 264] | 68.0 [4 to 483]
Bladder voiding efficiency (BVE) [Mean (Standard Deviation); unit: %] — Voided volume / (voided volume + post void residual): calculated from the voided volume measured by uroflowmetry and the post void residual measured by ultrasonography
  % | 58.38 (26.74) | 63.11 (24.13) | 59.82 (25.86)
Bladder voiding efficiency (BVE) [Median (Full Range); unit: %] — Voided volume / (voided volume + post void residual): calculated from the voided volume measured by uroflowmetry and the post void residual measured by ultrasonography
  % | 65.15 [0.6 to 88.6] | 73.46 [11.7 to 89.6] | 69.18 [0.6 to 89.6]
Bladder contractility index (BCI) (Only Male) [Mean (Standard Deviation); unit: Score on a scale] — Maximum detrusor pressure at peak urine flow (PdetQmax) + 5 × peak urine flow rate (Qmax): PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in men, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 150, normal 100-150, and weak < 100. No theoretical minimum and maximum value of the scale range exists. Population: This analysis was conducted only in male patients.
  Score on a scale
    number analyzed (Participants) | 27 | 11 | 38
    (all) | 64.604 (16.569) | 61.339 (16.629) | 63.659 (16.428)
Bladder contractility index (BCI) (Only Male) [Median (Full Range); unit: Score on a scale] — Maximum detrusor pressure at peak urine flow (PdetQmax) + 5 × peak urine flow rate (Qmax): PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in men, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 150, normal 100-150, and weak < 100. No theoretical minimum and maximum value of the scale range exists. Population: This analysis was conducted only in male patients.
  Score on a scale
    number analyzed (Participants) | 27 | 11 | 38
    (all) | 68.000 [13.77 to 98.00] | 60.000 [43.00 to 94.50] | 68.000 [13.77 to 98.00]
Projected isovolumetric pressure 1 (PIP1) (Only Female) [Mean (Standard Deviation); unit: Score on a scale] — PdetQmax + Qmax: PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in women, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 75, normal 30-75, and weak < 30. No theoretical minimum and maximum value of the scale range exists. Population: This analysis was conducted only in female patients.
  Score on a scale
    number analyzed (Participants) | 15 | 7 | 22
    (all) | 18.769 (6.591) | 20.561 (7.524) | 19.339 (6.773)
Projected isovolumetric pressure 1 (PIP1) (Only Female) [Median (Full Range); unit: Score on a scale] — PdetQmax + Qmax: PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in women, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 75, normal 30-75, and weak < 30. No theoretical minimum and maximum value of the scale range exists. Population: This analysis was conducted only in female patients.
  Score on a scale
    number analyzed (Participants) | 15 | 7 | 22
    (all) | 17.000 [8.50 to 32.40] | 21.000 [10.60 to 30.10] | 17.875 [8.50 to 32.40]

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Mean BCI for Male From Baseline to Week 12
Description: BCI indicates maxim um detrusor pressure at peak urine flow (PdetQmax) + 5 × peak urine flow rate (Qmax): PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in men, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 150, normal 100-150, and weak < 100. No theoretical minimum and maximum value of the scale range exists.
Time Frame: Baseline to Week 12
Population: PPS was used for the analysis. This analysis was conducted only in male patients in the PPS.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 27 | 11
Score on a scale
  BCI at baseline | 64.604 (16.569) | 61.339 (16.629)
  BCI at Week 12 | 75.156 (21.076) | 60.513 (16.708)
Statistical Analysis 1: Comparison: TAC-302; Baseline vs. Week 12 for the mean BCI in the TAC-302 group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 10.552, 95% CI 2-sided [5.514 to 15.590]
Statistical Analysis 2: Comparison: Placebo; Baseline vs. Week 12 for the mean BCI in the Placebo group; Test type: Superiority; p = 0.819, t-test, 2 sided; Mean Difference (Final Values) = -0.826, 95% CI 2-sided [-8.676 to 7.023]
Statistical Analysis 3: Comparison: TAC-302 vs Placebo; TAC-302 group vs. Placebo group for changes in the mean BCI from baseline to Week 12; Test type: Superiority; p = 0.015, t-test, 2 sided; Mean Difference (Final Values) = 11.378, 95% CI 2-sided [2.345 to 20.411], Standard Error of Mean 4.454

2. Primary Outcome: Changes in the Mean PIP1 for Female From Baseline to Week 12
Description: PIP1 indicates PdetQma x + Qmax: PdetQmax and Qmax denotes detrusor pressure at maximum flow and maximum flow rate in pressure flow study, respectively. This index is used to assess detrusor contractility in women, with a higher value indicating greater detrusor contractility. Contractility can be divided into strong > 75, normal 30-75, and weak < 30. No theoretical minimum and maximum value of the scale range exists.
Time Frame: Baseline to Week 12
Population: PPS was used for the analysis. This analysis was conducted only in female patients in the PPS.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 15 | 7
Score on a scale
  PIP1 at baseline | 18.769 (6.591) | 20.561 (7.524)
  PIP1 at Week 12 | 29.373 (9.369) | 25.487 (9.581)
Statistical Analysis 1: Comparison: TAC-302; Baseline vs. Week 12 for the mean PIP1 in the TAC-302 group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 10.604, 95% CI 2-sided [5.753 to 15.455], Standard Deviation 8.760
Statistical Analysis 2: Comparison: Placebo; Baseline vs. Week 12 for the mean PIP1 in the Placebo group; Test type: Superiority; p = 0.138, t-test, 2 sided; Mean Difference (Final Values) = 4.926, 95% CI 2-sided [-2.121 to 11.973], Standard Deviation 7.620
Statistical Analysis 3: Comparison: TAC-302 vs Placebo; TAC-302 group vs. Placebo group for changes in the mean PIP1 from baseline to Week 12; Test type: Superiority; p = 0.157, t-test, 2 sided; Mean Difference (Final Values) = 5.678, 95% CI 2-sided [-2.375 to 13.731], Standard Error of Mean 3.861

3. Secondary Outcome: Changes in the Mean BVE From Baseline to Week 12 (Overall)
Description: BVE indicates Voided volume / (voided volume + post void residual): calculated from the voided volume measured by uroflowmetry and the post void residual measured by ultrasonography.
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis. Therefore, the values presented here differ from those in the Baseline Characteristics module based on PPS.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
percentage
  BVE at baseline | 55.43 (26.82) | 63.71 (21.80)
  BVE at Week 12: number analyzed (Participants) | 48 | 23
  BVE at Week 12 | 66.79 (27.04) | 65.69 (28.98)
Statistical Analysis 1: Comparison: TAC-302; Baseline vs. Week 12 for the mean BVE in the TAC-302 group; Test type: Superiority; p = 0.006, t-test, 2 sided; Mean Difference (Final Values) = 10.91, 95% CI 2-sided [3.22 to 18.59], Standard Deviation 26.48
Statistical Analysis 2: Comparison: Placebo; Baseline vs. Week 12 for the mean BVE in the Placebo group; Test type: Superiority; p = 0.570, t-test, 2 sided; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [-6.27 to 11.10], Standard Deviation 20.09
Statistical Analysis 3: Comparison: TAC-302 vs Placebo; TAC-302 group vs. Placebo group for changes in the mean BVE from baseline to Week 12; Test type: Superiority; p = 0.178, t-test, 2 sided; Mean Difference (Final Values) = 8.49, 95% CI 2-sided [-3.96 to 20.95], Standard Error of Mean 6.24

4. Secondary Outcome: Changes in the Mean BVE From Baseline to Week 12 (In the Subgroup of Patients With Post Void Residual ≥ 50 mL at Baseline)
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis. Therefore, the values presented here differ from those in the Baseline Characteristics module based on PPS. This analysis was conducted in the subgroup of patients with post void residual ≥ 50 mL at baseline in the FAS.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 32 | 15
percentage
  BVE at baseline | 42.77 (24.66) | 55.95 (23.70)
  BVE at Week 12: number analyzed (Participants) | 29 | 15
  BVE at Week 12 | 61.66 (30.45) | 58.83 (26.15)
Statistical Analysis 1: Comparison: TAC-302; Baseline vs. Week 12 for the mean BVE in the TAC-302 group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 18.41, 95% CI 2-sided [9.13 to 27.69], Standard Deviation 24.39
Statistical Analysis 2: Comparison: Placebo; Baseline vs. Week 12 for the mean BVE in the Placebo group; Test type: Superiority; p = 0.489, t-test, 2 sided; Mean Difference (Final Values) = 2.88, 95% CI 2-sided [-5.81 to 11.58], Standard Deviation 15.70
Statistical Analysis 3: Comparison: TAC-302 vs Placebo; TAC-302 group vs. Placebo group for changes in the mean BVE from baseline to Week 12; Test type: Superiority; p = 0.031, t-test, 2 sided; Mean Difference (Final Values) = 15.53, 95% CI 2-sided [1.48 to 29.58], Standard Error of Mean 6.96

5. Secondary Outcome: Changes in the Mean BVE for Female From Baseline to Week 12 (In the Subgroup of Patients With Post Void Residual ≥ 100 mL at Baseline)
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis. Therefore, the values presented here differ from those in the Baseline Characteristics module based on PPS. This analysis was conducted In the subgroup of patients with post void residual ≥ 100 mL at baseline in the FAS.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 22 | 10
percentage
  BVE at baseline | 32.10 (20.16) | 44.03 (19.42)
  BVE at Week 12: number analyzed (Participants) | 19 | 10
  BVE at Week 12 | 54.71 (33.78) | 46.13 (18.72)
Statistical Analysis 1: Comparison: TAC-302; Baseline vs. Week 12 for the mean BVE in the TAC-302 group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 23.57, 95% CI 2-sided [11.26 to 35.88], Standard Deviation 25.54
Statistical Analysis 2: Comparison: Placebo; Baseline vs. Week 12 for the mean BVE in the Placebo group; Test type: Superiority; p = 0.708, t-test, 2 sided; Mean Difference (Final Values) = 2.10, 95% CI 2-sided [-10.19 to 14.40], Standard Deviation 17.18
Statistical Analysis 3: Comparison: TAC-302 vs Placebo; TAC-302 group vs. Placebo group for changes in the mean BVE from baseline to Week 12; Test type: Superiority; p = 0.025, t-test, 2 sided; Mean Difference (Final Values) = 21.47, 95% CI 2-sided [2.96 to 39.98], Standard Error of Mean 9.02

6. Secondary Outcome: Number of Micturitions Per 24 Hours at Baseline and Week 12
Description: On the basis of information from bladder diary records in the 3 days directly before each evaluation timepoint, an average of urinations per 24 hours was calculated. The patients with at least 8 urinations per 24 hours at registration were included in this study.
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis.
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Events
  Number of micturitions per 24 hours at baseline | 11.753 (3.065) | 11.764 (3.145)
  Number of micturitions per 24 hours at Week 12: number analyzed (Participants) | 49 | 23
  Number of micturitions per 24 hours at Week 12 | 10.830 (3.950) | 10.174 (2.348)

7. Secondary Outcome: Number of Urinary Urgency Episodes Per 24 Hours at Baseline and Week 12
Description: On the basis of information from bladder diary records in the 3 days directly before each evaluation timepoint, an average of urinary urgency episodes per 24 hours was calculated. The patients with at least one urinary urgency episode per 24 hours at registration were included in this study.
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis.
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Events
  Number of urinary urgency episodes per 24 hours at baseline | 5.452 (4.574) | 5.701 (3.878)
  Number of urinary urgency episodes per 24 hours at Week 12: number analyzed (Participants) | 49 | 23
  Number of urinary urgency episodes per 24 hours at Week 12 | 4.469 (6.095) | 2.493 (3.600)

8. Secondary Outcome: Overactive Bladder Symptom Score (OABSS) Total Score at Baseline and Week 12
Description: Overactive bladder symptoms were evaluated using the OABSS. The OABSS Total Score is the sum of four symptom scores: daytime frequency (score 0-2), nighttime frequency (score 0-3), urgency (score 0-5), and urgency incontinence (score 0-5). The range of scores is from 0 to 15 points with a higher score indicating greater severity. A score ≤ 5 was determined to be mild, a score of 6 to 11 was determined to be moderate and a score ≥ 12 was determined to be severe.
Time Frame: Baseline to Week 12
Population: FAS was used for the analysis.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
points
  OABSS total score at baseline | 8.7 (2.9) | 8.9 (2.4)
  OABSS total score at Week 12: number analyzed (Participants) | 49 | 23
  OABSS total score at Week 12 | 6.5 (3.2) | 7.3 (3.0)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: In tabulation of adverse events, the diagnoses entered on eCRFs were coded using the medical dictionary for regulatory activities (MedDRA) ver.22.1, and were presented as MedDRA preferred terms.
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: All treated patients in the treatment period were used for the analysis. This analysis set includes patients enrolled in the treatment period who took the investigational drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants
  Any adverse events | 24 | 9
  Deafness neurosensory | 0 | 1
  Constipation | 1 | 2
  Dental caries | 0 | 1
  Diarrhea | 2 | 0
  Diverticulum intestinal haemorrhagic | 0 | 1
  Glossitis | 0 | 1
  Haematochezia | 0 | 1
  Nausea | 0 | 1
  Vomiting | 0 | 1
  Pyrexia | 2 | 0
  Bacteriuria | 1 | 0
  Bronchitis | 1 | 1
  Cystitis | 1 | 1
  Gastroenteritis | 1 | 0
  Herpes virus infection | 0 | 1
  Influenza | 1 | 0
  Nasopharyngitis | 2 | 1
  Periodontitis | 0 | 1
  Pharyngitis | 1 | 1
  Pyuria | 2 | 0
  Urinary tract infection | 1 | 0
  Vulvitis | 1 | 0
  Enteritis infectious | 2 | 0
  Enterocolitis viral | 1 | 0
  Compression fracture | 1 | 0
  Fracture | 1 | 0
  Subdural haematoma | 1 | 0
  Contusion | 1 | 0
  Post procedural haematuria | 1 | 0
  Meniscus injury | 1 | 0
  Tooth dislocation | 1 | 0
  Blood creatinine phosphokinase increased | 1 | 0
  Back pain | 2 | 0
  Pain in extremity | 0 | 1
  Headache | 2 | 0
  Dysuria | 1 | 0
  Renal colic | 1 | 0
  Urethral pain | 1 | 0
  Prostatitis | 1 | 0
  Cough | 0 | 1
  Dermatitis contact | 0 | 1
  Miliaria | 1 | 0
  Rash | 0 | 1
  Orthostatic hypotension | 0 | 1

10. Secondary Outcome: Number of Participants With Adverse Drug Reactions
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: as for outcome 9
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants
  Any serious adverse events | 2 | 1
  Prostatitis | 1 | 0
  Subdural haematoma | 1 | 0
  Diverticulum intestinal haemorrhagic | 0 | 1

12. Secondary Outcome: Number of Participants With Adverse Events Leading to Death
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events Leading to Dose Discontinuation
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Adverse Events Leading to Dose Interruption
Description: as for outcome 9
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-302 | Placebo
Number analyzed (Participants) | 52 | 24
Participants
  Any adverse events leading to dose interruption | 2 | 1
  Enteritis infectious | 1 | 0
  Enterocolitis viral | 1 | 0
  Diverticulum intestinal haemorrhagic | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline to Week 13 (12 weeks in treatment period and 1 week in Follow-up period)
Description: All treated patients in the treatment period were used for the analysis. This analysis set includes patients enrolled in the treatment period who took the investigational drug at least once.
Arm/Group | TAC-302 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/52 | 1/24
Other Adverse Events (participants affected / at risk) | 24/52 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC-302 (N=52) | Placebo (N=24)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC-302 (N=52) | Placebo (N=24)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pyuria (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT03175029/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT03175029/SAP_001.pdf